CLINICAL TRIAL: NCT01039779
Title: A Randomized Trial of Tai Chi Exercise on Reducing Falls in Older Taiwanese People
Brief Title: Tai Chi Exercise in Older People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Collaborators: National Health Research Institutes, Taiwan (Other)
Responsible Party: Principal Investigator, Mau-Roung Lin, Professor, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NHRI-EX102-9805PI
Record Dates: First submitted 2009-12-24; First posted 2009-12-25 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Fallers Aged 60 Years and Older
Keywords: older fallers; tai chi
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lower-extremity exercise training (Active Comparator): This training will be tailored by physical therapists for each participant. A series of exercises will be applied to increase the stability of the trunk muscles and to strengthen the leg muscles.
  Interventions: Behavioral: Exercise
- Tai chi exercise (Active Comparator): Yang-style tai chi with 18 movements will be taught every week over the 6-month intervention period at a subject's residence by tai chi instructors
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Exercise will be taught every week over the 6-month intervention period at a subject's residence by instructors.

SUMMARY:
The effects of tai chi exercise and lower-extremity training on improving the primary outcome and secondary outcomes among older people will be compared.

DETAILED DESCRIPTION:
Does not desire.

ELIGIBILITY:
Inclusion Criteria:

* Persons aged 60 years and older and who require medical attention in the emergency rooms due to sustaining a fall.

Exclusion Criteria:

* A major unstable cardiopulmonary disease
* Cognitive impairment
* Contraindications to physical exercise
* The inability to ambulate
* Frail elderly.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 456 (Actual)
Dates: Start 2011-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
To ascertain the occurrence of falls | 18 months

SECONDARY OUTCOMES:
Fall-related outcomes of physical and psychological functions will assessed using direct interviews or performance tests at the subject's residence | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Mau-Roung Lin, Ph.D., Principal Investigator — Taipei Medical University
Locations (1):
- Taipei Medical University, Taipei, Taiwan